CLINICAL TRIAL: NCT01482962
Title: A Phase 3, Randomized, Two-Arm, Open-Label, Multicenter, International Trial of Alisertib (MLN8237) or Investigator's Choice (Selected Single Agent) in Patients With Relapsed or Refractory Peripheral T-Cell Lymphoma
Brief Title: Alisertib (MLN8237) or Investigator's Choice in Patients With Relapsed/Refractory Peripheral T-Cell Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C14012; 2011-003545-18 (EudraCT Number); DRKS00004503 (Registry Identifier: Germany (DRKS)); NL39566.068.12 (Registry Identifier: Netherlands (CCMO)); U1111-1181-8218 (Registry Identifier: WHO)
Record Dates: First submitted 2011-11-28; First posted 2011-12-01 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Relapsed Peripheral T-Cell Lymphoma; Refractory Peripheral T-Cell Lymphoma
Keywords: Drug Therapy
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — MLN 8237; 10-propargyl-10-deazaaminopterin; Gemcitabine; romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alisertib (Experimental): Alisertib 50 mg, enteric-coated tablet formulation, orally, twice daily for 7 consecutive days (Cycle Days 1-7) in a 21-day cycle (Up to 148 Weeks).
  Interventions: Drug: Alisertib
- Pralatrexate, or Romidepsin, or Gemcitabine (Active Comparator): Pralatrexate 30 mg/m^2, intravenous (IV) push over 3 to 5 minutes, once weekly, for 6 weeks in 7-week cycles with concurrent vitamin B12 and folic acid supplementation. Cycles were repeated every 7-weeks provided the participant continued to benefit from and tolerate the therapy (Up to 115 Weeks), or Gemcitabine 1,000 mg/m^2 over 30 minutes, intravenously, on Days 1, 8, and 15 of a 28-day cycle until the absence of disease progression or unacceptable toxicity (Up to 32 Weeks), or Romidepsin 14 mg/m^2, intravenously over a 4-hour period, on Days 1, 8, and 15 of a 28-cycle. Cycles were repeated every 28 days provided the patient continued to benefit from and tolerate the therapy (Up to 30 Weeks).
  Interventions: Drug: Pralatrexate; Drug: Gemcitabine; Drug: Romidepsin

INTERVENTIONS:
Drug: Alisertib — Alisertib enteric coated tablets
  Arms: Alisertib
Drug: Pralatrexate — Pralatrexate IV infusion
  Arms: Pralatrexate, or Romidepsin, or Gemcitabine
Drug: Gemcitabine — Gemcitabine IV infusion
  Arms: Pralatrexate, or Romidepsin, or Gemcitabine
Drug: Romidepsin — Romidepsin IV infusion
  Arms: Pralatrexate, or Romidepsin, or Gemcitabine

SUMMARY:
This is a phase 3, randomized, 2-arm, open-label, international trial evaluating alisertib compared with single-agent treatment, as selected by the investigator from the offered options of pralatrexate or gemcitabine or romidepsin, in participants with relapsed or refractory peripheral T-cell lymphoma (PTCL). Note: romidepsin was not used as a single-agent comparator outside the United States of America (USA) as supply was not available.

DETAILED DESCRIPTION:
The drug being tested in this study was Alisertib. Alisertib was tested to treat people who have relapsed/refractory peripheral T-cell lymphoma (PTCL).

This study evaluated alisertib for the improvement in overall response rate (ORR) compared with single-agent treatment, as selected by the investigator from the offered options of pralatrexate, romidepsin (US only), or gemcitabine, in participants with relapsed or refractory PTCL.

The study enrolled 271 patients. Participants were randomized (1:1) to one of 2 treatment arms:

* Alisertib
* Investigator's choice (Pralatrexate, Romidepsin, or Gemcitabine)

This multi-center trial was conducted worldwide. The overall time to participate in this study was approximately 5 years. Participants made multiple visits to the clinic, and then were contacted by telephone up to 42-months after the last participant was randomized, or until death, for follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants age 18 or older
* Participants with Peripheral T cell lymphoma (PTCL) (selected subtypes) according to World Health Organization (WHO) criteria and have relapsed or are refractory to at least 1 prior systemic, cytotoxic therapy for PTCL. Participants must have received conventional therapy as a prior therapy. Cutaneous-only disease is not permitted. Participants must have documented evidence of progressive and measurable disease.
* Tumor biopsy available for central hematopathologic review
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Female participants who are post menopausal for at least 1 year, surgically sterile, or agree to practice 2 effective methods of contraception through 30 days after the last dose of study drug or agree to abstain from heterosexual intercourse.
* Male participants who agree to practice effective barrier contraception through 6 months after the last dose of alisertib or agree to abstain from heterosexual intercourse
* Suitable venous access
* Voluntary written consent

Exclusion Criteria

* Known central nervous system lymphoma
* Systemic antineoplastic therapy, immunotherapy, investigational agent or radiation therapy within 4 weeks of first dose of study treatment or concomitant use during study
* Prior administration of an Aurora A kinase-targeted agent, including alisertib; or all of the 3 comparator drugs (pralatrexate, or romidepsin or gemcitabine; or known hypersensitivity)
* History of uncontrolled sleep apnea syndrome or other conditions that could result in excessive daytime sleepiness
* Cardiac condition as specified in study protocol, including left ventricular ejection fraction (LVEF) <40%
* Concomitant use of other medicines as specified in study protocol
* Participants with abnormal gastric or bowel function who require continuous treatment with H2-receptor antagonists or proton pump inhibitors
* Known active infection with human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C
* Autologous stem cell transplant less than 3 months prior to enrollment
* Participants who have undergone allogeneic stem cell or organ transplantation any time
* Inadequate blood levels, bone marrow or other organ function as specified in study protocol
* The participant must have recovered to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade ≤ 1 toxicity, to participant's baseline status (except alopecia), or deemed irreversible from the effects of prior cancer therapy
* Major surgery, serious infection, or infection requiring systemic antibiotic therapy within 14 days prior to the first dose of study treatment
* Female participants who are breastfeeding or pregnant
* Coexistent second malignancy or history of prior solid organ malignancy within previous 3 years
* Serious medical or psychiatric illness or laboratory abnormality that could, in the investigator's opinion, potentially interfere with the completion of treatment according to the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2012-06-11 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2017-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Takeda Oncology
Locations (151):
- United States (24):
  - Birmingham, Alabama
  - La Jolla, California
  - Orlando, Florida
  - Tampa, Florida
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Boston, Massachusetts
  - Detroit, Michigan
  - Rochester, Minnesota
  - Jefferson City, Missouri
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - Hackensack, New Jersey
  - Buffalo, New York
  - New York, New York
  - Syracuse, New York
  - Durham, North Carolina
  - Columbus, Ohio
  - Toledo, Ohio
  - Charleston, South Carolina
  - Houston, Texas
  - Burlington, Vermont
  - Seattle, Washington
  - Morgantown, West Virginia
- Australia (5):
  - Adelaide
  - Concord
  - Gosford
  - Hobart
  - St Leonards
- Austria (4):
  - Graz
  - Innsbruck
  - Salzburg
  - Vienna
- Belarus (2):
  - Minsk Didtrict
  - Vitebsk
- Belgium (6):
  - Bruges
  - Brussels
  - Ghent
  - Kortrijk
  - Turnhout
  - Yvoir
- Brazil (11):
  - Belo Horizonte
  - Campianas
  - Caxias do Sul
  - Curitiba
  - Goiânia
  - Porto Alegre
  - Porto Alegre/rs
  - Rio de Janeiro
  - Salvador
  - SAO Paulo - SP
  - São Paulo
- Bulgaria (3):
  - Pleven
  - Sofia
  - Varna
- Canada (2):
  - Ottawa, Ontario
  - Toronto, Ontario
- Chile (2):
  - Concepción
  - Santiago
- Prague, Czechia
- Denmark (2):
  - Arhus C
  - København Ø
- Egypt (4):
  - Alexandria
  - BENI SWEF
  - Cairo
  - Dakahlia
- France (6):
  - Bordeaux
  - Marseille
  - Paris
  - Pessac
  - Pierre-Bénite
  - Tours
- Germany (8):
  - Berlin
  - Essen
  - Freiburg im Breisgau
  - Göttingen
  - Homburg/saar
  - Mainz
  - München
  - Ulm
- Hungary (4):
  - Budapest
  - Debrecen
  - Kaposvár
  - Pécs
- Israel (6):
  - Beersheba
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Italy (10):
  - Bari
  - Bologna
  - Cagliari
  - Florence
  - Meldola
  - Modena
  - Ravenna
  - Rimini
  - Roma
  - Torino
- Mexico (5):
  - Durango Durango
  - México
  - Monterrey
  - Monterrey Nuevo LEON
  - San Luis Potosí City
- Netherlands (2):
  - Maastricht
  - Nieuwegein
- New Zealand (3):
  - Auckland
  - Christchurch
  - Takapuna
- Peru (2):
  - Arequipa
  - Lima
- Poland (6):
  - Bydgoszcz
  - Chorzów
  - Krakow
  - Lodz
  - Warsaw
  - Wroclaw
- Portugal (3):
  - Braga
  - Coimbra
  - Porto
- San Juan, PR, Puerto Rico
- Bucharest, Romania
- Russia (4):
  - Chelyabinsk
  - Moscow
  - Petrozavodsk
  - Saint Petersburg
- Slovakia (2):
  - Bratislava
  - Martin
- Spain (7):
  - Barcelona
  - Girona
  - Madrid
  - Pamplona
  - Salamanca
  - Seville
  - Valencia
- Sweden (3):
  - Linköping
  - Lund
  - Solna
- Turkey (Türkiye) (5):
  - Ankara
  - Denizli
  - Istanbul
  - Kayseri
  - Samsun
- United Kingdom (7):
  - Birmingham
  - Cardiff
  - Liverpool
  - Manchester
  - Newcastle upon Tyne
  - Southampton
  - Truro

REFERENCES:
- [Derived] O'Connor OA, Ozcan M, Jacobsen ED, Roncero JM, Trotman J, Demeter J, Masszi T, Pereira J, Ramchandren R, Beaven A, Caballero D, Horwitz SM, Lennard A, Turgut M, Hamerschlak N, d'Amore FA, Foss F, Kim WS, Leonard JP, Zinzani PL, Chiattone CS, Hsi ED, Trumper L, Liu H, Sheldon-Waniga E, Ullmann CD, Venkatakrishnan K, Leonard EJ, Shustov AR; Lumiere Study Investigators. Randomized Phase III Study of Alisertib or Investigator's Choice (Selected Single Agent) in Patients With Relapsed or Refractory Peripheral T-Cell Lymphoma. J Clin Oncol. 2019 Mar 10;37(8):613-623. doi: 10.1200/JCO.18.00899. Epub 2019 Feb 1. PMID 30707661

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 105 investigative sites in the United States including Puerto Rico, Canada, European Union, Russian Federation, Turkey, Israel, Australia, New Zealand and Latin America from 11 June 2012 to the end of study on 18 December 2017.
Pre-assignment Details: Participants with a diagnosis of Relapsed or Refractory Peripheral T-Cell Lymphoma were randomized 1:1 to either alisertib or comparator (investigator's choice of pralatrexate, romidepsin [USA only], or gemcitabine).
Period: Overall Study
Arm/Group | Alisertib | Pralatrexate, or Romidepsin, or Gemcitabine
Started | 138 | 133
Safety Population: Received Study Drug | 137 | 127
Completed | 0 | 0
Not Completed | 138 | 133
Not completed — Progressive Disease | 65 | 53
Not completed — Unsatisfactory Therapeutic Response | 37 | 23
Not completed — Adverse Event | 18 | 22
Not completed — Withdrawal by Participant | 8 | 13
Not completed — Hematopoietic Stem Cell Transplant | 3 | 9
Not completed — Other Reason | 1 | 5
Not completed — Study Terminated by Sponsor | 5 | 2
Not completed — Did not Receive Study Drug | 1 | 6

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population was defined as all participants who were randomized. The participants were analyzed according to the treatment they were randomized to receive, regardless of any errors of dosing.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alisertib | Pralatrexate, or Romidepsin, or Gemcitabine | Total
Number analyzed (Participants) | 138 | 133 | 271
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (12.69) | 61.4 (13.16) | 61.3 (12.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 47 | 93
  Male | 92 | 86 | 178
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 21 | 46
  Not Hispanic or Latino | 105 | 107 | 212
  Unknown or Not Reported | 8 | 5 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  White | 115 | 114 | 229
  Black or African American | 8 | 8 | 16
  Asian | 3 | 2 | 5
  Other | 7 | 7 | 14
  Not Reported | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  Australia | 5 | 4 | 9
  Austria | 2 | 2 | 4
  Belgium | 5 | 3 | 8
  Brazil | 12 | 10 | 22
  Bulgaria | 0 | 1 | 1
  Canada | 3 | 0 | 3
  Czech Republic | 5 | 2 | 7
  Denmark | 3 | 2 | 5
  France | 5 | 3 | 8
  Germany | 6 | 1 | 7
  Hungary | 9 | 7 | 16
  Israel | 0 | 3 | 3
  Italy | 6 | 6 | 12
  Mexico | 3 | 1 | 4
  Netherlands | 0 | 1 | 1
  New Zealand | 3 | 2 | 5
  Peru | 1 | 3 | 4
  Poland | 7 | 3 | 10
  Portugal | 1 | 1 | 2
  Puerto Rico | 0 | 1 | 1
  Romania | 2 | 1 | 3
  Russia | 4 | 4 | 8
  Spain | 14 | 11 | 25
  Sweden | 0 | 3 | 3
  Turkey | 10 | 11 | 21
  United Kingdom | 3 | 8 | 11
  United States | 29 | 39 | 68
Height [Mean (Standard Deviation); unit: cm] | 170.3 (9.80) | 168.2 (8.99) | 169.3 (9.45)
Weight [Mean (Standard Deviation); unit: kg] | 76.85 (17.242) | 74.63 (19.601) | 75.76 (18.437)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] — Population: Body surface area (m^2)=square root [height (cm)*weight (kg)/3600].
  m^2 | 1.897 (0.2465) | 1.855 (0.2562) | 1.877 (0.2517)

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Based on Independent Review Committee (IRC) Assessment
Description: ORR was defined as the percentage of participants who achieve Complete Response (CR) or Partial Response (PR) as assessed by the IRC using International Working Group (IWG) criteria. CR=Disappearance of all evidence of disease and PR=Regression of measurable disease and no new sites.
Time Frame: Every 8 weeks from date of first dose treatment; every 12 weeks after 40 week assessment; at end of treatment visit until progressive disease. Duration is approximately 3 years
Population: Response-evaluable population, participants with peripheral T-cell lymphoma confirmed by an independent hematopathology central review, with measurable disease at Baseline, who received at least 1 dose of alisertib or comparator and had postbaseline response assessment of CR, PR, stable disease (SD) or progressive disease (PD) by the IRC.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alisertib | Pralatrexate, or Romidepsin, or Gemcitabine
Number analyzed (Participants) | 102 | 92
percentage of participants | 33 [24 to 43] | 45 [34 to 55]
Statistical Analysis 1: Comparison: Alisertib vs Pralatrexate, or Romidepsin, or Gemcitabine; Test type: Superiority; p = 0.038, Cochran-Mantel-Haenszel — P-value was stratified using disease type, International Prognostic Index (IPI) Score and region as stratification factors; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.33 to 1.08]

2. Primary Outcome: Progression-Free Survival (PFS) Based on IRC Assessment
Description: PFS was defined as the time from the date of randomization to the date of first documentation of progressive disease (PD) or death due to any cause, whichever occurred first.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alisertib | Pralatrexate, or Romidepsin, or Gemcitabine
Number analyzed (Participants) | 138 | 133
days | 115 [83 to 174] | 104 [61 to 114]
Statistical Analysis 1: Comparison: Alisertib vs Pralatrexate, or Romidepsin, or Gemcitabine; Test type: Superiority; p = 0.177, Stratified Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.637 to 1.178] — Hazard ratio (HR) was based on a stratified Cox's proportional hazard regression model with stratification factors: disease type, IPI Score and region with treatment as a factor in the model

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death. Participants without documentation of death were censored at the date last known to be alive.
Time Frame: Participants were followed for survival for 2 years from date of last participant off study treatment, or death, whichever occurs first. Contacts were every 4 months (Median follow-up 519 days in the alisertib arm and 586 days in the comparative arm)
Population: ITT population was defined as all participants who were randomized. The participants were analyzed according to the treatment they were randomized to receive, regardless of any errors of dosing.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alisertib | Pralatrexate, or Romidepsin, or Gemcitabine
Number analyzed (Participants) | 138 | 133
days | 415 [263 to 514] | 367 [258 to 572]
Statistical Analysis 1: Comparison: Alisertib vs Pralatrexate, or Romidepsin, or Gemcitabine; Test type: Superiority; p = 0.338, Stratified Log-rank Test; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.707 to 1.369] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. A SAE is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/ birth defect or is a medically important event.
Time Frame: First dose to 30 days after last dose of study drug or comparator (Up to 152 Weeks)
Population: Safety population was defined as all participants who received at least 1 dose of alisertib, or one of the comparator drugs. Participants were analyzed according to the treatment actually received.
Measure: Number; unit: participants
Arm/Group | Alisertib | Pralatrexate, or Romidepsin, or Gemcitabine
Number analyzed (Participants) | 137 | 127
participants
  TEAE | 136 | 126
  SAE | 75 | 69

5. Secondary Outcome: Number of Participants With Clinically Important Abnormal Laboratory Values Reported as AEs
Description: Clinical laboratory tests included chemistry, hematology and urinalysis test. Clinically significant treatment-emergent laboratory abnormalities were reported by the investigator as TEAEs.
Time Frame: First dose to 30 days after last dose of study drug or comparator (Up to 152 Weeks)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Alisertib | Pralatrexate, or Romidepsin, or Gemcitabine
Number analyzed (Participants) | 137 | 127
participants
  Neutrophil Count Decreased | 18 | 14
  White Blood Cell Count Decreased | 17 | 10
  Lymphocyte Count Decreased | 6 | 5
  Monocyte Count Decreased | 2 | 1
  Lymphocyte Count Increased | 1 | 0
  Monocyte Count Increased | 1 | 0
  White Blood Cell Count Increased | 1 | 0
  Platelet Count Decreased | 15 | 22
  Alanine Aminotransferase Increased | 8 | 11
  Aspartate Aminotransferase Increased | 5 | 11
  Gamma-glutamyltransferase Increased | 6 | 3
  Blood Bilirubin Increased | 2 | 1
  Hepatic Enzyme Increased | 2 | 0
  Liver Function Test Abnormal | 0 | 1
  Transaminases Increased | 0 | 1
  Blood Alkaline Phosphatase Increased | 9 | 7
  Blood Lactate Dehydrogenase Increased | 5 | 1
  Blood Creatinine Increased | 3 | 7
  Blood Creatinine Decreased | 0 | 1
  Blood Urea Increased | 1 | 0
  Blood Potassium Decreased | 1 | 4
  Blood Magnesium Decreased | 1 | 2
  Blood Bicarbonate Decreased | 0 | 1
  Blood Calcium Decreased | 0 | 1
  Blood Calcium Increased | 1 | 0
  Blood Phosphorus Decreased | 0 | 1
  Calcium Ionised Increased | 1 | 0
  Haemoglobin Decreased | 1 | 3
  Haematocrit Increased | 1 | 2
  Haematocrit Decreased | 1 | 0
  Coagulation Factor XIII Level Decreased | 1 | 0
  International Normalised Ratio Increased | 1 | 0
  Blood Albumin Decreased | 0 | 2
  Myocardial Necrosis Marker Increased | 1 | 0
  Troponin Increased | 0 | 1
  Blood Glucose Increased | 0 | 1
  Immunoglobulins Increased | 1 | 0
  Blood Uric Acid Increased | 1 | 0
  Enterovirus Test Positive | 0 | 1

6. Secondary Outcome: Number of Participants With Clinically Important Vital Sign Measurements Reported as AEs
Description: Vital signs included blood pressure, heart rate and temperature. Individual clinically significant changes in vital signs were reported by the investigator as TEAEs.
Time Frame: First dose to 30 days after last dose of study drug or comparator (Up to 152 Weeks)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Alisertib | Pralatrexate, or Romidepsin, or Gemcitabine
Number analyzed (Participants) | 137 | 127
participants
  Heart Rate Increased | 1 | 0
  Body Temperature Increased | 0 | 1
  Hypotension | 4 | 6
  Orthostatic Hypotension | 2 | 1
  Hypertension | 5 | 7
  Pyrexia | 48 | 40

7. Secondary Outcome: Complete Response (CR) Rate
Description: Complete Response (CR) rate is defined as the percentage of participants with CR as assessed by the IRC using IWG criteria (2007 Cheson). CR= Disappearance of all evidence of disease.
Time Frame: At the end of every 8 weeks from date of first dose treatment; every 12 weeks after 40 week assessment; at end of treatment visit until PD (approximately 3 years)
Population: Response-evaluable population was defined as participants with peripheral T-cell lymphoma confirmed by an independent hematopathology central review, with measurable disease at baseline, who receive at least 1 dose of alisertib or the comparator drug, and 1 postbaseline response assessment of CR, PR, SD or PD by the independent radiology committee.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alisertib | Pralatrexate, or Romidepsin, or Gemcitabine
Number analyzed (Participants) | 102 | 92
percentage of participants | 18 [11 to 26] | 27 [18 to 37]

8. Secondary Outcome: Time to Disease Progression (TTP)
Description: Time to Progression (TTP) was defined as the time from the date of randomization to the date of first documentation of PD/relapse.
Time Frame: At the end of every 8 weeks from date of first dose treatment; every 12 weeks after 40 week assessment; at end of treatment visit until progressive disease. Duration is approximately 3 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alisertib | Pralatrexate, or Romidepsin, or Gemcitabine
Number analyzed (Participants) | 138 | 133
days | 162 [114 to 231] | 116 [101 to 227]
Statistical Analysis 1: Comparison: Alisertib vs Pralatrexate, or Romidepsin, or Gemcitabine; Test type: Superiority; p = 0.362, Stratified Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.679 to 1.329] — Hazard ratio was based on a stratified Cox's proportional hazard regression model with stratification factors: disease type, IPI Score and region with treatment as a factor in the model

9. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the date of first documentation of a PR or better to the date of first documentation of progressive disease (PD)/relapse for responders as assessed by the IRC using IWG criteria. Responders without documentation of PD/relapse were censored at the date of last response assessment that was stable disease (SD) or better.
Time Frame: as for outcome 8
Population: All responders in response-evaluable population defined as participants with peripheral T-cell lymphoma confirmed by independent hematopathology central review with measurable disease at baseline who receive at least 1 dose of alisertib or comparator drug and 1 postbaseline response assessment of CR, PR, SD or PD by independent radiology committee.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alisertib | Pralatrexate, or Romidepsin, or Gemcitabine
Number analyzed (Participants) | 34 | 41
days | 225 [125 to NA] — Upper Limit Confidence Interval was not estimable due to the insufficient number of participants with the event. | 172 [119 to NA] — Upper Limit Confidence Interval was not estimable due to the insufficient number of participants with the event.

10. Secondary Outcome: Time to Response
Description: Time to Response is defined as the time from the date of randomization to the date of first documentation of PR or better.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alisertib | Pralatrexate, or Romidepsin, or Gemcitabine
Number analyzed (Participants) | 34 | 41
days | 62 [57 to 67] | 64 [60 to 71]

11. Secondary Outcome: Time to Subsequent Antineoplastic Therapy
Description: Time to subsequent antineoplastic therapy was defined as the time from randomization to the first date of subsequent antineoplastic therapy (excluding transplant). Participants without subsequent antineoplastic therapy were censored at the date of death or last known to be alive.
Time Frame: From date of last study drug to date of subsequent antineoplastic therapy, if required; approximately 3 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alisertib | Pralatrexate, or Romidepsin, or Gemcitabine
Number analyzed (Participants) | 138 | 133
days | 336 [201 to 490] | 233 [144 to 429]

12. Secondary Outcome: Plasma Concentration-time Data to Contribute to Future Population Pharmacokinetics (PK) Analysis
Time Frame: Cycle 1, Days 1 and 7; Cycle 2, Day 8; Cycle 3, Day 8; Cycle 4, Day 8. Duration is approximately 4 months.
Population: This Outcome Measure was registered in error and is not a Primary or Secondary Outcome Measure.
Arm/Group | Alisertib
Number analyzed (Participants) | 0

13. Secondary Outcome: Change Form Baseline in Reported Symptoms and Quality of Life (QoL) Assessment Per Functional Assessment of Cancer Therapy-Lymphoma (FACT-LYM) for Functioning and Symptoms
Description: The FACT-LYM includes the Functional Assessment of Cancer Therapy General Scale (FACT-G) and a 15-item lymphoma-specific subscale (LYM) over the past week. The FACT-G has 27 items that incorporate 4 scales including physical well-being (PWB; 7 items), social/family well-being (SWB, 7 items), emotional well-being (EWB; 6 items), and functional well-being (FWB; 7 items). The combined FACT-LYM instrument consists of a total of a 42 item questionnaire. Each question is answered on a 5- point scale of 0 (not at all) to 4 (very much) for a total possible score of 168. Higher scores indicate better well-being and a positive change from Baseline indicates improvement.
Time Frame: Baseline and End of Treatment (EOT) (Up to 152 Weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alisertib | Pralatrexate, or Romidepsin, or Gemcitabine
Number analyzed (Participants) | 138 | 133
score on a scale
  Physical Well-Being, EOT: number analyzed (Participants) | 81 | 70
  Physical Well-Being, EOT | -2.4 (6.21) | -1.3 (5.27)
  Social/Family Well-Being, EOT: number analyzed (Participants) | 81 | 69
  Social/Family Well-Being, EOT | -0.3 (4.50) | 0.0 (4.44)
  Emotional Well-Being, EOT: number analyzed (Participants) | 80 | 67
  Emotional Well-Being, EOT | -1.4 (4.59) | -0.8 (3.93)
  Functional Well-Being, EOT: number analyzed (Participants) | 80 | 66
  Functional Well-Being, EOT | -2.4 (5.40) | -0.3 (4.79)

ADVERSE EVENTS:
Time Frame: First dose to 30 days after last dose of study drug or comparator (Up to 152 Weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Adverse events for arm "Gemcitabine or Pralatrexate or Romidepsin" were reported separately for each treatment received and reported as Gemcitabine, Pralatrexate, and Romidepsin.
Groups:
- Gemcitabine: Gemcitabine 1,000 mg/m^2 over 30 minutes, intravenously, on Days 1, 8, and 15 of a 28-day cycle until the absence of disease progression or unacceptable toxicity (Up to 32 Weeks).
- Pralatrexate: Pralatrexate 30 mg/m^2, intravenous (IV) push over 3 to 5 minutes, once weekly, for 6 weeks in 7-week cycles with concurrent vitamin B12 and folic acid supplementation. Cycles were repeated every 7-weeks provided the participant continued to benefit from and tolerate the therapy (Up to 115 Weeks).
- Romidepsin: Romidepsin 14 mg/m^2, intravenously over a 4-hour period, on Days 1, 8, and 15 of a 28-cycle. Cycles were repeated every 28 days provided the patient continued to benefit from and tolerate the therapy (Up to 30 Weeks).
Arm/Group | Alisertib | Gemcitabine | Pralatrexate | Romidepsin
All-Cause Mortality (participants affected / at risk) | 11/137 | 5/29 | 8/76 | 2/22
Serious Adverse Events (participants affected / at risk) | 75/137 | 18/29 | 46/76 | 6/22
Other Adverse Events (participants affected / at risk) | 134/137 | 29/29 | 72/76 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib (N=137) | Gemcitabine (N=29) | Pralatrexate (N=76) | Romidepsin (N=22)
Pneumonia (Infections and infestations) | 9 | 0 | 4 | 0 — One treatment-emergent death occurred during treatment with alisertib and is related.
Lung infection (Infections and infestations) | 1 | 1 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 2 | 0 | 2 | 0 — One treatment-emergent death occurred during treatment with alisertib and is not related.
Septic shock (Infections and infestations) | 4 | 0 | 1 | 0 — Four treatment-emergent deaths occurred during treatment with alisertib, two related and two not related.
Skin infection (Infections and infestations) | 1 | 0 | 2 | 0 — One treatment-emergent death occurred during treatment with pralatrexate and is not related.
Dermatitis infected (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Epiglottitis (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 1 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 2 | 0
Erysipelas (Infections and infestations) | 2 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 1 | 0 | 0
Oral infection (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia haemophilus (Infections and infestations) | 1 | 0 | 0 | 0
Eczema herpeticum (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 24 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 1 | 4 | 0
Anaemia (Blood and lymphatic system disorders) | 7 | 0 | 2 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 12 | 6 | 6 | 1
General physical health deterioration (General disorders) | 1 | 0 | 3 | 0 — Three treatment-emergent deaths occurred during treatment with pralatrexate and are not related.
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 1 | 0 — Two treatment-emergent deaths occurred during treatment, one with alisertib, not related and one with pralatrexate, related.
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 1
Hypothermia (General disorders) | 1 | 0 | 0 | 0
Catheter site phlebitis (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0
Adverse drug reaction (General disorders) | 0 | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with gemcitabine and is related.
Stomatitis (Gastrointestinal disorders) | 7 | 0 | 11 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with gemcitabine and is not related.
Jejunal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with pralatrexate and is not related.
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 — Two treatment-emergent deaths occurred during treatment, one with alisertib and one with pralatrexate and are not related.
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 — One treatment-emergent death occurred during treatment with gemcitabine and is not related.
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with pralatrexate and is not related.
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Peripheral T-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1 | 2 — Five treatment-emergent deaths occurred during treatment and are not related, two with alisertib, one with gemcitabine, and two with romidepsin.
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with alisertib and is not related.
Anaplastic large cell lymphoma T- and null-cell types (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with gemcitabine and is not related.
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0 | 0
Carotid artery aneurysm (Nervous system disorders) | 0 | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 2 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Anaphylactoid reaction (Immune system disorders) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Adult T-cell lymphoma/leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib (N=137) | Gemcitabine (N=29) | Pralatrexate (N=76) | Romidepsin (N=22)
Diarrhoea (Gastrointestinal disorders) | 61 | 5 | 18 | 10
Stomatitis (Gastrointestinal disorders) | 42 | 0 | 48 | 2
Nausea (Gastrointestinal disorders) | 35 | 7 | 23 | 15
Constipation (Gastrointestinal disorders) | 17 | 6 | 20 | 3
Vomiting (Gastrointestinal disorders) | 18 | 3 | 15 | 4
Abdominal pain (Gastrointestinal disorders) | 16 | 1 | 7 | 2
Dyspepsia (Gastrointestinal disorders) | 12 | 1 | 5 | 2
Abdominal pain upper (Gastrointestinal disorders) | 8 | 2 | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 5 | 0 | 5 | 0
Odynophagia (Gastrointestinal disorders) | 2 | 0 | 5 | 0
Anaemia (Blood and lymphatic system disorders) | 74 | 7 | 30 | 6
Neutropenia (Blood and lymphatic system disorders) | 66 | 11 | 21 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 51 | 12 | 29 | 7
Leukopenia (Blood and lymphatic system disorders) | 39 | 6 | 6 | 2
Lymphopenia (Blood and lymphatic system disorders) | 14 | 2 | 5 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 1 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0
Fatigue (General disorders) | 49 | 11 | 14 | 6
Pyrexia (General disorders) | 42 | 7 | 20 | 3
Oedema peripheral (General disorders) | 21 | 5 | 10 | 5
Asthenia (General disorders) | 24 | 2 | 10 | 0
Chills (General disorders) | 9 | 2 | 5 | 2
Malaise (General disorders) | 4 | 3 | 1 | 1
Mucosal inflammation (General disorders) | 3 | 1 | 5 | 0
Peripheral swelling (General disorders) | 1 | 2 | 2 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 2
Platelet count decreased (Investigations) | 16 | 11 | 6 | 5
Neutrophil count decreased (Investigations) | 18 | 5 | 5 | 4
White blood cell count decreased (Investigations) | 16 | 5 | 3 | 2
Alanine aminotransferase increased (Investigations) | 8 | 2 | 9 | 0
Weight decreased (Investigations) | 12 | 1 | 6 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 3 | 8 | 0
Blood alkaline phosphatase increased (Investigations) | 9 | 1 | 5 | 1
Blood creatinine increased (Investigations) | 3 | 3 | 3 | 2
Haemoglobin decreased (Investigations) | 1 | 2 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 43 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 1 | 11 | 5
Rash (Skin and subcutaneous tissue disorders) | 5 | 1 | 7 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 5 | 2 | 4 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 2 | 4 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 0 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 4 | 17 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 4 | 8 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 11 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 6 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 4 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 14 | 3 | 3 | 1
Influenza (Infections and infestations) | 8 | 1 | 3 | 0
Conjunctivitis (Infections and infestations) | 4 | 0 | 7 | 0
Pneumonia (Infections and infestations) | 4 | 0 | 5 | 1
Sinusitis (Infections and infestations) | 5 | 0 | 2 | 3
Viral upper respiratory tract infection (Infections and infestations) | 4 | 2 | 3 | 1
Skin infection (Infections and infestations) | 2 | 1 | 6 | 0
Bronchitis (Infections and infestations) | 4 | 0 | 4 | 0
Pharyngitis (Infections and infestations) | 3 | 0 | 4 | 0
Oral herpes (Infections and infestations) | 3 | 3 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 27 | 1 | 14 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 0 | 5 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 | 1 | 6 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 7 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 4 | 1
Dizziness (Nervous system disorders) | 16 | 2 | 6 | 1
Headache (Nervous system disorders) | 15 | 2 | 5 | 2
Somnolence (Nervous system disorders) | 15 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 3 | 0 | 2 | 4
Disturbance in attention (Nervous system disorders) | 2 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 3 | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 0 | 6 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 1 | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 2 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 12 | 2 | 3 | 1
Anxiety (Psychiatric disorders) | 5 | 1 | 4 | 3
Hypertension (Vascular disorders) | 5 | 2 | 2 | 3
Hypotension (Vascular disorders) | 4 | 2 | 2 | 2
Tachycardia (Cardiac disorders) | 5 | 0 | 4 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 2
Palpitations (Cardiac disorders) | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.